CLINICAL TRIAL: NCT03671161
Title: Combination of Flash Glucose Measure System and Continuous Subcutaneous Insulin Infusion Therapy in Patients With Type 1 Diabetes and Poor Glycemic Control Related to Very Few Self-blood Glucose Measurements
Brief Title: Flash Glucose Measure System and Continuous Subcutaneous Insulin Infusion Therapy in Poorly Controlled Diabetes Type 1 Patients
Acronym: FREESTYLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CIC1421-18-15
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Diabetes Mellitus, Type 1
Keywords: Diabetes Type 1; Insulin Pump; flash glucose monitoring; hypoglycemia; ketoacidocetosis; DTSQ; HFS
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: 19 patients with type 1 diabetes, HbA1c >9% (75 mmol/mol), multi daily insulin injections ( MDI) and who perform less than 2 SMBG /day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with poorly controlled diabetes type 1 (Experimental): Adults with type 1 diabetes, HbA1c >9% (75 mmol/mol), multi daily insulin injections ( MDI) and who perform less than 2 SMBG /day swithced to Insulin Pump and flash glucose monitoring
  Interventions: Device: Insulin Pump and flash glucose monitoring

INTERVENTIONS:
Device: Insulin Pump and flash glucose monitoring — Adults with type 1 diabetes, HbA1c >9% (75 mmol/mol), multi daily insulin injections ( MDI) and who perform less than 2 SMBG /day. Patients will be switched to insulin pump and start a FGM system (Free Style Libre®) during 6 months.

SUMMARY:
Patients with diabetes type 1 with poor glycemic control will be switched to insulin pump and FGM system (Flash Glucose Monitoring) during 6 months, correlated to the hypothesis that they could benefit from this intervention by being reengaged in diabetes self-management.

DETAILED DESCRIPTION:
This is a non-controlled proof of concept prospective pilot study in adults with type 1 diabetes, HbA1c >9% (75 mmol/mol), multi daily insulin injections ( MDI) and who perform less than 2 SMBG /day. Patients will be switched to insulin pump and started a FGM system (Free Style Libre®) during 6 months, hoping this intervention can reengage patients in self-management, reduce HbA1c without increasing the risk of ketoacidocetosis (DKA) and severe hypoglycemia (SH), and keep the DTSQ (Diabetes Treatment Satisfaction Questionnaire) and HFS (Hypoglycemia Fear Scale) at good levels.

ELIGIBILITY:
Inclusion Criteria:

* adults with type 1 diabetes, aged between 18 and 55, HbA1c >9% (75 mmol/mol), multi daily insulin injections (MDI) treatment, maximum 2 SMBG /day

Exclusion Criteria:

* diabetes with less than 1 year duration, severe active retinopathy requiring laser therapy, severe psychiatric illness, pregnancy, inability to communicate in French, concomitant severe active disease, patients already using a FGM or a CGM

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c ≥1% | 6 months
  Blood samples at baseline and 6 months
Number of severe hypoglycemia episodes | 6 months
  Number of severe hypoglycemia episodes, evaluated by flash glucose monitoring
Number of ketoacidosis episodes | 6 months

SECONDARY OUTCOMES:
Any positive change in DTSQ scale (ΔDTSQM6-DTSQM0>0) (Diabetes Treatment Satisfaction Questionnaire) | 6 months
  Filling questionnaires at baseline and 6 months. DTSQ (Diabetes treatment questionnaire) includes 8 items, each score from 0 to 6 with a higher score indicating better outcome
Any positive change in HFS scale (Hypoglycemia Fear Scale) | 6 months
  Filling questionnaires at baseline and 6 months. HFS (Hypoglycemia fear scale) assesses participant's fear of hypoglycemia both overall and separately for behavior (10 items) and worry (17 items), both items scoring from 1 to 5, with lower score indicating better outcome
Number of Hypoglycemia episodes | 6 months
  Number of hypoglycemia episodes, evaluated by Flash glucose monitoring
Frequency of hypoglycemia episodes | 6 months
  Frequency of hypoglycemia episodes, evaluated by Flash glucose monitoring
Frequency of severe hypoglycemia episodes | 6 months
  Frequency of severe hypoglycemia episodes, evaluated by Flash glucose monitoring
Frequency of ketoacidosis episodes | 6 months
Any changes in Weight | 6 months
  Weight measures at baseline 2 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Halbron M, Bourron O, Andreelli F, Ciangura C, Jacqueminet S, Popelier M, Bosquet F, Rouanet S, Amouyal C, Hartemann A. Insulin Pump Combined with Flash Glucose Monitoring: A Therapeutic Option to Improve Glycemic Control in Severely Nonadherent Patients with Type 1 Diabetes. Diabetes Technol Ther. 2019 Jul;21(7):409-412. doi: 10.1089/dia.2019.0041. PMID 31265349